CLINICAL TRIAL: NCT00407030
Title: Prospective, Double-blind, Placebo-controlled, Randomized, Multi-center Trial With a Double-blind Parallel-group Extension Period to Investigate the Efficacy and Safety of Different Doses of IncobotulinumtoxinA (Xeomin) in the Treatment of Cervical Dystonia
Brief Title: IncobotulinumtoxinA (Xeomin) Versus Placebo in the Treatment of Cervical Dystonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 60201-0408
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2010-12-31 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- incobotulinumtoxinA (Xeomin) (240 Units) (Experimental): incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), 240 units, total volume 4.8mL; Mode of administration: intramuscular injection
  Interventions: Drug: incobotulinumtoxinA (Xeomin) (240 Units)
- incobotulinumtoxinA (Xeomin) (120 Units) (Experimental): incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), 120 units, total volume 4.8 mL; Mode of administration: intramuscular injection
  Interventions: Drug: incobotulinumtoxinA (Xeomin) (120 Units)
- Placebo (Placebo Comparator): Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection Dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl, corresponding total placebo volume 4.8 mL; Mode of administration: intramuscular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: incobotulinumtoxinA (Xeomin) (240 Units) — incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (240 Units)
  Arms: incobotulinumtoxinA (Xeomin) (240 Units)
Drug: incobotulinumtoxinA (Xeomin) (120 Units) — incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (120 Units)
  Arms: incobotulinumtoxinA (Xeomin) (120 Units)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
At baseline patients received incobotulinumtoxinA (Xeomin) or placebo. Thereafter, all patients who entered the extension period were treated with up to five injection sessions of incobotulinumtoxinA (Xeomin) during the extension period.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female outpatients between ages 18 and 75 years inclusive)
* A clinical diagnosis of cervical dystonia (i.e. spasmodic torticollis) with predominantly rotational form and a need for injection (determined by the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) -Total score)
* TWSTRS-Total score >= 20
* TWSTRS-Severity score >= 10
* TWSTRS-Disability score >= 3
* TWSTRS-Pain score >= 1
* On a stable dose of medications (if any) used for focal dystonia treatment (e.g. anticholinergics and benzodiazepines) for at least 3 months prior to and expected throughout the Main Period
* For pre-treated patients only: Source documentation of the last two consecutive injection sessions with Botulinum Toxin and stable therapeutic response directly prior to trial entry
* For pre-treated patients only: At least 10 weeks must have been passed between the last injection with Botulinum Toxin for cervical dystonia and baseline
* For pre-treated patients only: The most recent injection with Botulinum Toxin must have been maximal 300 Units of type A or 12,000 Units of type B

Main Exclusion Criteria:

* Traumatic torticollis or tardive torticollis
* TWSTRS-Severity score for anterocollis >= 2 points (pure anterocollis)
* TWSTRS-Severity score for retrocollis >= 2 points (pure retrocollis)
* Myotomy or denervation surgery in the affected muscles (e.g. peripheral denervation and/or spinal cord stimulation)
* Hypersensitivity to human serum albumin, sucrose, or Botulinum Toxin Type A
* Diagnosis of myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant neuromuscular disease which might interfere with the trial
* Current swallowing disorder of any origin (dysphagia scale >= 3, i.e. severe, with swallowing difficulties and requiring a change in diet)
* Marked limitation on passive range of motion that suggests contractures or other structural abnormality, e.g. cervical contractures or cervical spine syndrome
* Treatment with Botulinum Toxins for any indication other than cervical dystonia within 4 months prior to baseline and during the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2006-07; Primary Completion 2008-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Comella, M.D., Study Chair — Rush University Medical Center, 1725 West Harrison Street, Suite 755, Chicago, 60612 Illinois, USA
Locations (1):
- Dallas, Texas, United States

REFERENCES:
- [Result] Comella CL, Jankovic J, Truong DD, Hanschmann A, Grafe S; U.S. XEOMIN Cervical Dystonia Study Group. Efficacy and safety of incobotulinumtoxinA (NT 201, XEOMIN(R), botulinum neurotoxin type A, without accessory proteins) in patients with cervical dystonia. J Neurol Sci. 2011 Sep 15;308(1-2):103-9. doi: 10.1016/j.jns.2011.05.041. Epub 2011 Jul 18. PMID 21764407
- [Result] Evidente VG, Fernandez HH, LeDoux MS, Brashear A, Grafe S, Hanschmann A, Comella CL. A randomized, double-blind study of repeated incobotulinumtoxinA (Xeomin((R))) in cervical dystonia. J Neural Transm (Vienna). 2013 Dec;120(12):1699-707. doi: 10.1007/s00702-013-1048-3. Epub 2013 Jun 19. PMID 23779062

RESULTS

PARTICIPANT FLOW:
Groups:
- incobotulinumtoxinA (Xeomin) (240 Units): incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kD), free from complexing proteins")(active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection, 240 units; Mode of administration: intramuscular injection
- incobotulinumtoxinA (Xeomin) (120 Units): incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kD), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection, 120 units; Mode of administration: intramuscular injection
- Placebo: Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection Dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl; Mode of administration: intramuscular injection
Period: Main Period - 8 to 20 Weeks
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Started | 81 | 78 | 74
Completed | 76 | 75 | 68
Not Completed | 5 | 3 | 6
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Consent Withdrawn | 1 | 1 | 1
Not completed — Withdrawal Criteria Occurred | 0 | 0 | 1
Not completed — Patient Decision | 1 | 0 | 0
Period: Extension Period - up to 68 Weeks
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Started | 111 (2 subjects did not enter the Ext. Period, 3 subjects never expressed any need for a new injection) | 103 (2 subjects did not enter the Ext. Period, 3 subjects never expressed any need for a new injection) | 0 (After the Main Period all patients were randomly assigned to the 2 active treatment arms.)
Completed | 84 | 74 | 0
Not Completed | 27 | 29 | 0
Not completed — Withdrawal Criteria Occurred | 4 | 5 | 0
Not completed — Lack of Efficacy | 11 | 11 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Consent Withdrawn | 4 | 4 | 0
Not completed — Lost to Follow-up | 5 | 5 | 0
Not completed — Patient Decision | 1 | 2 | 0
Not completed — Physician Decision | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo | Total
Number analyzed (Participants) | 81 | 78 | 74 | 233
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (12.2) | 52.8 (11.5) | 52.4 (10.8) | 52.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 51 | 49 | 154
  Male | 27 | 27 | 25 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) -Total Score at Week 4 After Injection of the Main Period - Xeomin (240 Units) Versus Placebo
Description: The TWSTRS-Total score is the sum of scores of the three components of the scale:
  * TWSTRS-Severity score which ranges from 0 (=absence of severity) to 35 points (=maximum severity)
  * TWSTRS-Pain score which ranges from 0 (=no pain) to 20 (=maximum pain)
  * TWSTRS-Disability score which ranges from 0 (=no disability) to 30 (=maximum disability).
  The TWSTRS total score ranges from 0 (=best value) to 85 (=worst value). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, week 4
Population: Intention to treat population: all participants randomized were included in the primary efficacy analysis; missing values were imputed using the worst case strategy, i.e. imputation by baseline value
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | Placebo
Number analyzed (Participants) | 81 | 74
points on a scale | -7.3 (2.18) | 1.6 (2.28)
Statistical Analysis 1: Comparison: incobotulinumtoxinA (Xeomin) (240 Units) vs Placebo; Hierarchical testing: Primary null hypothesis: incobotulinumtoxinA (Xeomin) (240 Units) identical to placebo. Rejection of 1st hypothesis lead to test of 2nd null hypothesis: incobotulinumtoxinA (Xeomin) (120 Units) identical to placebo. Rejection of 2nd hypothesis lead to test of 3rd null hypothesis: incobotulinumtoxinA (Xeomin) (240 Units) identical to incobotulinumtoxinA (Xeomin) (120 Units). 3 separate models were used to test these hypotheses which results in different LS means estimates; Test type: Superiority or Other; p < 0.001, ANCOVA — Due to the hierarchical testing no adjustment of type I error was necessary; Independent variables in the model were treatment, baseline TWSTRS-Total score, gender, age, pre-treatment of cervical dystonia, and pooled center; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-12.0 to -5.9]

2. Secondary Outcome: Change From Baseline in the TWSTRS-Total Score
Description: as for outcome 1
Time Frame: Baseline, week 8, final visit (up to 20 weeks after injection of the Main Period)
Population: Intention to treat population with missing values imputed using the worst case strategy, i.e. imputation by baseline value
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Number analyzed (Participants) | 81 | 78 | 74
points on a scale
  Baseline - Week 8 | -8.2 (10.54) | -6.9 (11.15) | 0.4 (7.17)
  Baseline - Final Visit | -4.6 (7.52) | -3.6 (8.07) | 1.7 (6.15)

3. Secondary Outcome: Change From Baseline in the TWSTRS Disability Subscore
Description: TWSTRS-Disability score which ranges from 0 (=no disability)to 30 (=maximum disability). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, week 4, week 8, final visit (up to 20 weeks after injection of the Main Period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Number analyzed (Participants) | 81 | 78 | 74
points on a scale
  Baseline - Week 4 | -3.0 (4.35) | -3.3 (4.72) | 0.0 (3.41)
  Baseline - Week 8 | -2.4 (3.98) | -2.1 (4.86) | 0.8 (3.27)
  Baseline - Final Visit | -1.3 (3.13) | -1.4 (3.82) | 1.0 (3.32)

4. Secondary Outcome: Change From Baseline in the TWSTRS Severity Subscore
Description: TWSTRS-Severity score which ranges from 0 (=absence of severity) to 35 points (=maximum severity). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, week 4, week 8, final visit (up to 20 weeks after injection of the Main Period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Number analyzed (Participants) | 81 | 78 | 74
points on a scale
  Baseline - Week 4 | -5.5 (5.99) | -3.9 (4.34) | -1.9 (3.96)
  Baseline - Week 8 | -3.5 (5.39) | -3.1 (4.39) | -0.9 (3.57)
  Baseline - Final Visit | -1.9 (3.83) | -1.1 (3.18) | -0.2 (3.07)

5. Secondary Outcome: Change From Baseline in the TWSTRS Pain Subscore
Description: TWSTRS-Pain score which ranges from 0 (=no pain) to 20 (=maximum pain). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, week 4, week 8, final visit (up to 20 weeks after injection of the Main Period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Number analyzed (Participants) | 81 | 78 | 74
points on a scale
  Baseline - Week 4 | -2.4 (4.36) | -2.7 (4.55) | -0.3 (2.97)
  Baseline - Week 8 | -2.3 (4.32) | -1.8 (4.15) | 0.6 (2.82)
  Baseline - Final Visit | -1.3 (3.40) | -1.1 (3.96) | 0.9 (2.56)

6. Secondary Outcome: Patient Evaluation of Global Response (PEGR) at Final Visit
Description: The PEGR is a descriptive subjective 9-point response scale ranging from "complete abolishment of signs and symptoms" (value=+4) down to "very marked worsening" (value=-4).
Time Frame: Final visit (up to 20 weeks after injection of the Main Period)
Population: Intention to treat population with missing values imputed by "no effect"
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Number analyzed (Participants) | 81 | 78 | 74
points on a scale | 1.3 (1.84) | 1.3 (1.77) | -0.2 (1.34)

7. Primary Outcome: Change From Baseline in the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) -Total Score at Week 4 After Injection of the Main Period - Xeomin (120 Units) Versus Placebo
Description: as for outcome 1
Time Frame: Baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Number analyzed (Participants) | 78 | 74
points on a scale | -10.8 (2.11) | -3.3 (2.20)
Statistical Analysis 1: Comparison: incobotulinumtoxinA (Xeomin) (120 Units) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Due to the hierarchical testing no adjustment of type I error was necessary; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-10.4 to -4.6]

8. Primary Outcome: Change From Baseline in the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) -Total Score at Week 4 After Injection of the Main Period - Xeomin (240 Units) Versus Xeomin (120 Units)
Description: as for outcome 1
Time Frame: Baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units)
Number analyzed (Participants) | 81 | 78
points on a scale | -10.5 (2.25) | -9.2 (2.27)
Statistical Analysis 1: Comparison: incobotulinumtoxinA (Xeomin) (240 Units) vs incobotulinumtoxinA (Xeomin) (120 Units); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.447, ANCOVA — Due to the hierarchical testing no adjustment of type I error was necessary; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.1 to 4.6]

ADVERSE EVENTS:
Time Frame: All SAEs/AEs during Double-Blind Period after Injection, i.e. up to 8-20 weeks after Main Period injection.
Description: The table of "Other Adverse Events" includes all non-serious AEs. Only results and AEs of the Double-Blind Period are given as the Extension Period was not placebo-controlled. The investigator asked the patient for AEs systematically at each visit.
Arm/Group | incobotulinumtoxinA (Xeomin) (240 Units) | incobotulinumtoxinA (Xeomin) (120 Units) | Placebo
Serious Adverse Events (participants affected / at risk) | 4/81 | 0/78 | 0/74
Other Adverse Events (participants affected / at risk) | 27/81 | 26/78 | 14/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | incobotulinumtoxinA (Xeomin) (240 Units) (N=81) | incobotulinumtoxinA (Xeomin) (120 Units) (N=78) | Placebo (N=74)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | incobotulinumtoxinA (Xeomin) (240 Units) (N=81) | incobotulinumtoxinA (Xeomin) (120 Units) (N=78) | Placebo (N=74)
Dysphagia (Gastrointestinal disorders) | 15 (17) | 9 (10) | 2 (2)
Injection site pain (General disorders) | 3 (3) | 7 (7) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (12) | 5 (5) | 1 (1)
Musculosceletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (8) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 4 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results to be published without written agreement by sponsor; manuscripts to be sent to sponsor at least 6 weeks before submission. Sponsor to give written opinion within 30 days. Sponsor is entitled to exert influence on the contents of publications, to postpone publications up to 36 months after end of the study, and to name co-authors. In case of justified doubts of sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.